CLINICAL TRIAL: NCT02485808
Title: Symptoms of Lower Urinary Tract Dysfunction Research Network (LURN) Phenotyping Study Protocol
Brief Title: Symptoms of Lower Urinary Tract Dysfunction Phenotyping Study
Status: Completed | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other); Northwestern University (Other); Duke University (Other); University of Iowa (Other); University of Washington (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: LURN Phenotyping Study V8.0; U01DK100017 (NIH); U01DK100011 (NIH); U01DK099932 (NIH); U01DK099879 (NIH); U01DK097780 (NIH); U01DK097779 (NIH); U01DK097776 (NIH); U01DK097772 (NIH)
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower Urinary Tract Symptoms; Bladder Symptoms; Overactive Bladder; Urinary Urgency; Lower Urinary Tract Dysfunction
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Overactive | interventions — Magnetic Resonance Spectroscopy; Pain Threshold

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood - DNA Plasma Urine Vaginal Cultures (women) Perineal Cultures (men) Saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Surgical: Men and women presenting for clinical care for whom surgical treatment of their lower urinary symptoms is planned.
  There will be no interventions, as this is an observational cohort.
  Interventions: Other: None-observational
- Medical: Men and women presenting for clinical care for whom medical treatment of their lower urinary symptoms is planned.
  There will be no interventions, as this is an observational cohort.
  Interventions: Other: None-observational
- Controls: Men and women who are not experiencing lower urinary tract symptoms.
  This group will undergo MRI, pain and auditory sensitivity testing.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Other: Multimodal Automated Sensory Testing System; Other: Auditory Sensitivity Test
- Neuroimaging & Sensory Testing: Subjects from the Medical and Surgical Cohorts who agree to additional testing in the form of neuroimaging (via fMRI) and multimodal sensory testing.
  This group will undergo MRI, pain and auditory sensitivity testing.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Other: Multimodal Automated Sensory Testing System; Other: Auditory Sensitivity Test

INTERVENTIONS:
Other: None-observational — For surgical patients, follow-up assessments will occur 3 and 12 months after the surgery. For medical patients, follow-up assessments will occur 3 and 12 months after the baseline assessment.
  Groups: Medical; Surgical
Procedure: Magnetic Resonance Imaging (MRI) — One time MRI scanning session examining brain structure and function in a resting state and after water consumption.
  Other Names: MRI
  Groups: Controls; Neuroimaging & Sensory Testing
Other: Multimodal Automated Sensory Testing System — Pressure pain thresholds will be assess using computer-controlled pressures delivered by a device called the Multimodal Automated Sensory Testing System (MAST) device on to the subjects thumbnail bed.
  Other Names: Pain Sensitivity
  Groups: Controls; Neuroimaging & Sensory Testing
Other: Auditory Sensitivity Test — Subjects' sensitivity to sound will be evaluated using a series of sounds delivered by a standard audiometer device.
  Groups: Controls; Neuroimaging & Sensory Testing

SUMMARY:
The purpose of this study is to advance our understanding of people who experience urinary and bladder problems. We are interested in learning about people's experiences with urinary symptoms and how these symptoms will be managed. We want to understand the important differences among people and what factors affect urinary and bladder problems. After all of the information is collected, we will have a better understanding of how to improve the care and treatment for people who have urinary and bladder problems.

DETAILED DESCRIPTION:
The Symptoms of Lower Urinary Tract Dysfunction Research Network (LURN) was established by the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) to advance our understanding of lower urinary tract dysfunction (LUTD) in women and men. LUTD is a term intended to be comprehensive and to challenge current paradigms about how symptomatic pelvic disorders are defined as 'diseases.' Lower urinary tract symptoms (LUTS) are likely caused and exacerbated by a variety of factors and thus do not represent the manifestation of a single disease. Clinical management of LUTD, including treatment outcomes, remains suboptimal since the biological and psychosocial factors that initiate, exacerbate, and modify this group of symptoms remain largely unknown. As an initial effort to better characterize the biological and psychosocial factors that initiate, exacerbate, and modify LUTS, the LURN investigators will establish a prospective Observational Cohort Study of men and women with LUTS presenting for the first time to LURN physicians.

Information to be obtained from study participants initially (at time of enrollment) includes a standardized clinical examination, medical history, select testing of the lower urinary tract, and participants' self-report of LUTS, pelvic floor symptoms including sexual function and bowel symptoms, depression, anxiety, sleep patterns, stress, metabolic risk factors, and health-related quality of life. We will also collect serum, urine, saliva, and perineal swabs from men and vaginal swabs from women for storage at the NIDDK Sample Repository for future study by the LURN investigators and the broader research community. This information will be used to construct subgroups of patients who have similar symptoms, clinical presentations, comorbidities, pelvic floor dysfunctions, and psychological profiles. These patient characteristics and behaviors likely affect the evaluation, diagnosis, and/or treatment of LUTS. Additional information will be collected 3 months and 12 months after enrollment or 3 and 12 months after surgery for patients receiving surgical treatment, and will include an interval clinical history, participants' self-report of LUTS, pelvic floor symptoms including sexual function and bowel symptoms, depression, anxiety, and health-related quality of life. We will also collect biological samples at 3 and 12 months after enrollment.

The LURN Neuroimaging and Sensory Testing component of the study will investigate abnormal sensation of the lower urinary tract at the level of the organism. Subjects and controls will have a one-time visit soon after their baseline visit, where they will undergo an fMRI scan of their brain and multimodal quantitative sensory testing assessing perceptual responses to physical stimuli (pain and sound).

The information to be collected from the prospective Observational Cohort Study will be limited and not sufficient to fully understand the pathophysiology and biology of LUTS. Therefore, the Observational Cohort Study will serve as the basis for further LURN studies. The long-term goal of the LURN is to better characterize patients with LUTD in order to advance future research on the pathophysiology of these

ELIGIBILITY:
Inclusion Criteria:

1. Men and women presenting for new patient visits for evaluation or treatment of LUTS to one of the LURN physicians.
2. Age ≥ 18 years.
3. The presence of any of the symptoms reported in Table 1, based on responses to the LUTS Tool with a one month recall period.
4. The ability to give informed consent and complete self-reported questionnaires electronically.

Table 1: LUTS Appropriate for Study Inclusion

* Daytime frequency
* Nocturia
* Urgency
* Incontinence/leakage (various types)
* Poor or absent sensation of bladder filling
* Slow/weak stream
* Splitting or spraying
* Intermittent stream/Double voiding
* Hesitancy
* Straining
* Dribbling at the end of flow
* Paruesis (shy bladder syndrome)
* Poor or absent sensation of urethra during void
* Feeling of incomplete emptying
* Post-micturition dribble (delayed)
* Abnormal bladder or urethral sensations

Exclusion Criteria:

1. Gross hematuria.
2. Significant neurologic disease or injury, including but not limited to: cerebral vascular accident with residual defect, Alzheimer's dementia, Parkinson's disease, traumatic brain injury, spinal cord injury, complicated spinal surgery, multiple sclerosis.
3. Primary complaint is pelvic pain.
4. Diagnosis of interstitial cystitis, chronic prostatitis, or chronic orchialgia.
5. Pelvic or endoscopic GU surgery within the preceding 6 months (not including diagnostic cystoscopy).
6. Current sexually transmitted infection. (deferral; subject can enroll after negative culture)
7. Ongoing symptomatic urethral stricture.
8. History of lower urinary tract or pelvic malignancy.
9. Current chemotherapy or other cancer therapy.
10. Pelvic device or implant complication (e.g., sling or mesh complications).
11. Current functioning neurostimulator.
12. Botox injection to the bladder or pelvic structures within the preceding 12 months.
13. In men, prostate biopsy in the previous 3 months.
14. In women, pregnancy.
15. History of cystitis caused by tuberculosis, radiation therapy, or Cytoxan/cyclophosphamide therapy.
16. Augmentation cystoplasty or cystectomy.
17. Presence of urinary tract fistula.
18. Current major psychiatric disorder or other psychiatric or medical issues that would interfere with study participation (e.g., dementia, psychosis, etc.).
19. Inability to relay valid information, actively participate in the study, or provide informed consent (includes uncontrolled psychiatric disease).
20. Difficulty reading or communicating in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New patients with LUTS presenting to LURN clinical sites will be screened for participation based on the inclusion and exclusion criteria (below).
Sampling Method: Non-Probability Sample
Enrollment: 1879 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Clinically relevant subgroups of patients with lower urinary tract symptoms | Baseline
  Identification of patient clusters based on their symptoms, clinical assessments, and/or other characteristics.

SECONDARY OUTCOMES:
Change in lower urinary tract symptoms | baseline, 3 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Weinfurt, PhD, Study Chair — Duke University; Claire Yang, MD, Study Chair — University of Washington; Robert M Merion, MD, FACS, Principal Investigator — Arbor Research Collaborative for Health - DCC
Locations (6):
- United States (6):
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
We do not plan to make IPD available.

REFERENCES:
- [Background] Coyne KS, Matza LS, Kopp ZS, Thompson C, Henry D, Irwin DE, Artibani W, Herschorn S, Milsom I. Examining lower urinary tract symptom constellations using cluster analysis. BJU Int. 2008 May;101(10):1267-73. doi: 10.1111/j.1464-410X.2008.07598.x. Epub 2008 Mar 11. PMID 18336611
- [Background] Coyne KS, Barsdorf AI, Thompson C, Ireland A, Milsom I, Chapple C, Kopp ZS, Bavendam T. Moving towards a comprehensive assessment of lower urinary tract symptoms (LUTS). Neurourol Urodyn. 2012 Apr;31(4):448-54. doi: 10.1002/nau.21202. Epub 2012 Mar 6. PMID 22396308
- [Background] Bower WF, Yip SK, Yeung CK. Dysfunctional elimination symptoms in childhood and adulthood. J Urol. 2005 Oct;174(4 Pt 2):1623-7; discussion 1627-8. doi: 10.1097/01.ju.0000176599.91836.12. PMID 16148668
- [Derived] Helmuth ME, Smith AR, Glaser AP, Yang CC, Cameron AP, Henry Lai H, Griffith JW, Eric Jelovsek J, Quentin Clemens J, Helfand BT, Merion RM, Andreev VP; and the LURN Study Group. Phenotyping Men With Lower Urinary Tract Symptoms: Results From the Symptoms of Lower Urinary Tract Dysfunction Research Network. Neurourol Urodyn. 2025 Jan;44(1):178-193. doi: 10.1002/nau.25596. Epub 2024 Oct 7. PMID 39370868
- [Derived] Lai HH, Rutlin J, Smith AR, Helmuth ME, Hokanson JA, Yang CC, Clemens JQ, Magnotta VA, Bretschneider CE, Kenton K, DeLancey JOL, John K, Kirkali Z, Shimony JS. Structural Changes in Brain White Matter Tracts Associated With Overactive Bladder Revealed by Diffusion Tensor Magnetic Resonance Imaging: Findings From a Symptoms of Lower Urinary Tract Dysfunction Research Network Cross-Sectional Case-Control Study. J Urol. 2024 Aug;212(2):351-361. doi: 10.1097/JU.0000000000004022. Epub 2024 May 8. PMID 38717915
- [Derived] Mawla I, Schrepf A, Kutch JJ, Helmuth ME, Smith AR, Ichesco E, Yang CC, Andreev VP, Kreder KJ, Bradley CS, Magnotta VA, Kirkali Z, Harris RE, Lai HH, Harte SE. Naturalistic Bladder Filling Reveals Subtypes in Overactive Bladder Syndrome That Differentially Engages Urinary Urgency-Related Brain Circuits: Results From the Symptoms of Lower Urinary Tract Dysfunction Research Network (LURN). J Urol. 2024 Jan;211(1):111-123. doi: 10.1097/JU.0000000000003699. Epub 2023 Oct 5. PMID 37796776
- [Derived] Harte SE, Wiseman J, Wang Y, Smith AR, Yang CC, Helmuth M, Kreder K, Kruger GH, Gillespie BW, Amundsen C, Kirkali Z, Lai HH; LURN Study Group. Experimental Pain and Auditory Sensitivity in Overactive Bladder Syndrome: A Symptoms of the Lower Urinary Tract Dysfunction Research Network (LURN) Study. J Urol. 2022 Jan;207(1):161-171. doi: 10.1097/JU.0000000000002147. Epub 2022 Aug 25. PMID 34428922
- [Derived] Helmuth ME, Smith AR, Andreev VP, Liu G; LURN Study Group; Lai HH, Cameron AP, Siddiqui NY. Use of Euclidean length to measure urinary incontinence severity based on the lower urinary tract symptoms tool. Am J Obstet Gynecol. 2018 Mar;218(3):357-359. doi: 10.1016/j.ajog.2017.12.219. Epub 2017 Dec 26. No abstract available. PMID 29288065
- See also: Study website — https://nih-lurn.org